CLINICAL TRIAL: NCT00103870
Title: Music Engagement for Non-Pharmacological Analgesia R21 AT001586-01
Brief Title: Mind Engagement With Music for Nondrug Pain Relief
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: David H. Bradshaw, PhD, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 12579; R21AT001586-01A1 (NIH)
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Pain
Keywords: Music Therapy; Electric Stimulation; Electric Shock; Analgesics; Distraction
MeSH Terms: conditions — Pain

INTERVENTIONS:
Procedure: Electrodermal stimulation
Procedure: Music listening task

SUMMARY:
The purpose of this study is to determine whether engaging in music listening tasks can reduce the perception of pain and provide nondrug pain relief.

Study hypotheses: 1) Performing a highly engaging listening task reduces psychophysiological arousal to painful stimuli. 2) Psychophysiological arousal to painful stimuli is a function of the complexity of the auditory signal. 3) Signal complexity and task difficulty interact to produce the greatest engagement and maximum reduction in psychophysiological arousal to painful stimuli.

DETAILED DESCRIPTION:
Music therapy involves the use of music to promote, maintain, and restore physical and mental health. Music analgesia is one aspect of music therapy focused on the reduction of pain through the use of musical activities. This study will build upon music analgesia data in the development of a new concept called music engagement. This concept is based on constructivist theory, which presumes that the brain continuously constructs and revises a model of reality. Pain is a constructed reality that may be prevented from being felt if a person is actively engaged in constructing another perceptual experience. Music listening is an activity that requires activation and integration of many complex cognitive and emotional processes; therefore, being actively engaged in music listening can impede the construction of pain if the listener can fully construct and sustain the music experience. This study will determine whether engagement in and construction of a music listening experience can reduce perceptions of pain.

This trial will comprise two studies and will require two days of participation. At study start, participants will have electrodes placed on a finger on their non-dominant hand and on other body parts to record skin conductance and electrical brain activity. Participants will also wear a headset to have their pupil movement measured. Tone synthesis software will be used to generate different tones. In Study 1, a familiar tune, selected by the participant, will be played against a background of varying tones. Occasionally, notes of the tune will be missing or displaced. Participants will be asked to identify the deviant notes while receiving painful fingertip shocks; they will be instructed to focus on the task and ignore the shocks. Study 1 will consist of three different conditions (easy, hard, and no condition). In the easy condition, the background tones occur far from the pitch range of the tune, making missing or displaced notes easy to detect. In the hard condition, the pitch range of the background tones will be adjacent to that of the tune, making the tune difficult to discern from the background tones. In the no task condition, participants will hear the familiar tune with random background tones, but they will be instructed to pay no attention to the tune or the tones.

Participants will report their pain experiences in both a retrospective report and a concurrent report. For the retrospective report, participants will report the highest, lowest, and average levels of pain experienced during the preceding block of trials. For the concurrent report, participants will give both a report of the level of pain experienced immediately following each shock episode. At each of the two sessions participants take part in, there will be two sets of trial blocks, one with pain reports and one without. There will be two blocks for each of the three music task conditions for a total of twelve blocks per session. Within each block, sixteen 7- to 11-second shocks will be given.

In Study 2, participants will take part in two types of listening tasks, one with only tones and one with both a tune and background tones. There will be three tasks in the tone condition (no task, easy task, and hard task). In the no task condition, participants will hear repeated tones; they will be instructed to pay no attention to the tones. In the easy condition, the deviant tones will be easily detectable; in the hard condition, they will be less detectable. During each condition, participants will receive painful fingertip shocks.

The second task condition is similar to Study 1; participants will listen to a familiar tune with various tones in the background. Participants will be given fingertip shocks and will be asked to identify deviant notes for both the easy and hard conditions. For the no task condition, participants will be instructed to pay no attention to the tune or background tones. Participants will not be required to report pain in this part of the study. Participants will receive two blocks of trials for each of the six task conditions. Fingertip shocks will vary in intensity with the interval between shocks varying between 7 and 11 seconds.

Pain self-reports (Study 1), deviant note detections, skin conductance, pupil dilation, and electroencephalogram changes following stimulations will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all study requirements

Exclusion Criteria:

* Abnormal hearing
* Severe allergies to skin preparations
* Psychoactive drugs
* Hypertension drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Reduction in psychophysiological markers for nociceptive responses

SECONDARY OUTCOMES:
Level of engagement as measured by engagement ratings and absorption scale

CONTACTS AND LOCATIONS:
Overall Officials: David H. Bradshaw, PhD, Principal Investigator — University of Utah Pain Research Center
Locations (1):
- University of Utah Pain Research Center, Salt Lake City, Utah, United States